CLINICAL TRIAL: NCT04831281
Title: A Randomized, Placebo-Controlled, Double-Blind Study of ATH-1017 Treatment in Subjects With Parkinson's Disease Dementia or Dementia With Lewy Bodies
Brief Title: ATH-1017 Treatment in Subjects With Parkinson's Disease Dementia or Dementia With Lewy Bodies (SHAPE Trial)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment ended early due to study design limitations.
Sponsor: Athira Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATH-1017-PD-0201
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease Dementia; Dementia With Lewy Bodies
Keywords: Parkinson's Disease Dementia; Dementia with Lewy Bodies; Dementia; HGF/MET; Hepatocyte Growth Factor; Neurotrophic; ATH-1017; Event-Related Potential; ERP P300
MeSH Terms: conditions — Lewy Body Disease; Dementia; Deafness, Autosomal Recessive 39

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 40mg Dose (Experimental): Daily subcutaneous injection of 40mg ATH-1017
  Interventions: Drug: ATH-1017
- 70mg Dose (Experimental): Daily subcutaneous injection of 70mg ATH-1017
  Interventions: Drug: ATH-1017
- Placebo (Placebo Comparator): Daily subcutaneous injection of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATH-1017 — Daily subcutaneous injection of ATH-1017 in a pre-filled syringe
  Arms: 40mg Dose; 70mg Dose
Drug: Placebo — Daily subcutaneous injection of Placebo in a pre-filled syringe
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety and treatment effects of fosgonimeton (ATH-1017) in subjects with Parkinson's Disease Dementia or Dementia with Lewy Bodies, with a randomized treatment duration of 26 weeks.

DETAILED DESCRIPTION:
The study is designed to evaluate the safety and treatment effects of ATH-1017 in subjects with Parkinson's Disease Dementia or Dementia with Lewy Bodies, with a randomized, double-blind, placebo-controlled, parallel-arm treatment duration of 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with confirmed diagnosis of Parkinson's disease or Dementia with Lewy Bodies
* MoCA score 11 to 23, inclusive, at screening
* Probable Parkinson's Disease Dementia or Lewy Body Dementia
* BMI between ≥ 16and ≤ 35 kg/m2 for females and between≥ 18 and ≤ 35 kg/m2 for males at Screening
* Reliable and capable support person/caregiver, who is willing to accept responsibility for supervising the treatment or, if required, administering study drug, and assessing the condition of the subject throughout the study in accordance with all protocol requirements

Exclusion Criteria:

* Hoehn-Yahr stage 5
* History of significant neurological disease other than PDD or DLB that may affect cognition at onset of dementia
* Subjects on deep brain stimulation
* History of brain MRI scan indicative of any other significant abnormality
* History of unexplained loss of consciousness, and epileptic fits
* Hearing test result considered unacceptable for auditory ERP P300 assessment
* Diagnosis of severe major depressive disorder even without psychotic features (GDS score [15-item scale] >7 at Screening)
* Significant suicide risk based on C-SSRS
* Significant psychosis (according to Diagnostic and Statistical Manual of Mental Disorders)
* Moderate or severe substance abuse disorder (according to DSM-5)
* Myocardial infarction or unstable angina within the last 6 months
* Clinically significant cardiac arrhythmia (including atrial fibrillation), cardiomyopathy, or cardiac conduction defect (note: pacemaker is acceptable)
* Clinically significant ECG abnormality at Screening
* Chronic kidney disease (eGFR < 45 mL/min using Cockcroft-Gault formula)
* Hepatic impairment with alanine aminotransferase or aspartate aminotransferase > 2 times the upper limit of normal, or Child-Pugh class B and C
* Malignant tumor within 3 years before Screening
* Memantine at any dose or combination
* Donepezil at 23 mg

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - QUEST Research Institute, Farmington Hills, Michigan
  - Summit Research Network, Portland, Oregon
  - Center for Cognitive Health, Portland, Oregon
  - Keystone Clinical Studies LLC, Plymouth Meeting, Pennsylvania
  - Northwest Clinical Research Center, Bellevue, Washington
  - Evergreen Health Research, Kirkland, Washington
  - Inland Northwest Research LLC, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a total of 7 centers in the United States (US).
Pre-assignment Details: This was a multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study comparing ATH-1017 40 milligrams per day (mg/day) and ATH-1017 70 mg/day with placebo in participants with Parkinson's Disease Dementia or Dementia with Lewy Bodies.
Groups:
- Placebo: Participants were randomized to receive placebo via subcutaneous (SC) injection once-daily (QD) preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
- ATH-1017 40 Milligrams (mg): Participants were randomized to receive ATH-1017 40mg via subcutaneous (SC) injection once-daily (QD) preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
- ATH-1017 70 mg: Participants were randomized to receive ATH-1017 70mg via subcutaneous (SC) injection once-daily (QD) preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
Period: Overall Study
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg) | ATH-1017 70 mg
Started | 9 | 9 | 10
Completed | 7 | 7 | 5
Not Completed | 2 | 2 | 5
Not completed — Adverse Event | 1 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Undetermined | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: included all randomized participants who received at least one dose of the study medication.
Groups:
- Placebo: Participants were randomized to receive placebo via subcutaneous (SC) injection QD preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
- ATH-1017 40 mg: Participants were randomized to receive ATH-1017 40 mg via subcutaneous (SC) injection QD preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
- ATH-1017 70 mg: Participants were randomized to receive ATH-1017 70 mg via subcutaneous (SC) injection QD preferably during daytime. The first SC injection of study drug was performed at site under supervision. The participant should withhold study drug administration on the day of subsequent clinic visits; study drug administration was done on site under supervision of site staff at these visits. Clinic visits took place on Day 1 and thereafter at Weeks 2, 6, 12, 16, 20, and 26, with a safety follow-up visit scheduled 4 weeks after completion of the double-blind period at Week 30
- Total: Total of all reporting groups
Arm/Group | Placebo | ATH-1017 40 mg | ATH-1017 70 mg | Total
Number analyzed (Participants) | 9 | 9 | 10 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (4.86) | 70.7 (9.89) | 74.2 (7.5) | 73.3 (7.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 7
  Male | 5 | 8 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 9 | 9 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 9 | 10 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Global Statistical Test (GST) Score at Baseline
Description: The Global Statistical Test (GST) score is a composite of the change from baseline (CFB) z-scores to Week 26 in the Alzheimer's Disease Assessment Scale - Cognitive Subscale, 13-Item Version (ADAS-Cog13; range 0-85; higher scores indicate greater impairment) and Event Related Potential P300 Latency (ERP P300; longer latency (milliseconds) indicates greater impairment). This composite approach was used to assess overall change in disease status and treatment effects of ATH-1017.
  The GST score was defined as a single outcome variable based on standardizing and combining individual patient-level z-score of change from baseline cognition (ADAS-Cog13) and ERP P300 latency scores. The between-group difference was calculated by subtracting the mean GST score for placebo from the mean GST score for ATH-1017. A negative value based on GST scores (ATH-1017 minus placebo) indicates a favorable response to ATH-1017, while a positive value favors placebo.
Time Frame: Baseline
Population: Modified intent to treat population.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Placebo | ATH-1017 40 mg | ATH-1017 70 mg
Number analyzed (Participants) | 9 | 7 | 9
Z-score | -0.222 (0.6365) | 0.332 (0.6337) | -0.036 (1.0050)

2. Secondary Outcome: Event-related Potential (ERP) P300 Latency at Baseline
Description: ERP P300 was a method of recording brain activity elicited by external stimuli, for example (e.g.), an oddball auditory stimulus, particularly of working memory access. The participant had to perform a task related to auditory stimuli in order to assess the P300 component (latency). The stimulus consisted of an oddball paradigm with 2 sound stimuli. Stimuli were presented through headphones and auditory stimulation for P300 was assessed in a recording lasting up to 10 minutes. It was calculated as the average across the pre-dose values at Baseline visit.
Time Frame: Baseline
Population: Modified intent to treat population.
Measure: Mean (Standard Deviation); unit: Millisecond (ms)
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg) | ATH-1017 70 mg
Number analyzed (Participants) | 9 | 7 | 9
Millisecond (ms) | 381.84 (51.739) | 373.19 (18.669) | 367.84 (45.635)

3. Secondary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog13) at Baseline
Description: The Alzheimer's Disease Assessment Scale - Cognitive Subscale, 13-Item Version (ADAS-Cog13) is designed to measure cognitive symptom change. The test comprises 9 performance items and 4 clinician-rated items (total score ranging from 0 to 85). Higher scores indicate more severe cognitive impairment.
Time Frame: Baseline
Population: Modified intent to treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg) | ATH-1017 70 mg
Number analyzed (Participants) | 9 | 7 | 9
score on a scale | 16.9 (6.94) | 29.7 (10.03) | 23.8 (11.49)

ADVERSE EVENTS:
Time Frame: Up to Week 30
Description: Safety population which included all randomized participants who received at least one dose of the study medication.
Arm/Group | Placebo | ATH-1017 40 Milligrams (mg) | ATH-1017 70 mg
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 1/10
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/9 | 1/10
Other Adverse Events (participants affected / at risk) | 7/9 | 9/9 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | ATH-1017 40 Milligrams (mg) (N=9) | ATH-1017 70 mg (N=10)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Psychotic symptom (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=9) | ATH-1017 40 Milligrams (mg) (N=9) | ATH-1017 70 mg (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 2 | 4
Injection site nodule (General disorders) | 0 | 3 | 2
Injection site pain (General disorders) | 0 | 1 | 2
Injection site pruritus (General disorders) | 0 | 1 | 1
Injection site warmth (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Injection site hypersensitivity (General disorders) | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Herpes pharyngitis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lip infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 4
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Freezing phenomenon (Nervous system disorders) | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0
Psychotic symptom (Psychiatric disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was stopped early prior to the accrual of the planned sample size of approximately 75 evaluable participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT04831281/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT04831281/SAP_001.pdf